CLINICAL TRIAL: NCT06175780
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of KY-0118 in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: Phase I Study of KY-0118 in Subjects With Locally Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Novatim Immune Therapeutics (Zhejiang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY-0118-ZJKY
Record Dates: First submitted 2023-11-29; First posted 2023-12-19 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Neoplasms; Neoplasms by Histologic Type
MeSH Terms: conditions — Neoplasms; Neoplasms by Histologic Type

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KY-0118 (Experimental)
  Interventions: Drug: KY-0118
- Cohort1: KY-0118 (Experimental)
  Interventions: Drug: KY-0118
- Cohort2: KY-0118 (Experimental)
  Interventions: Drug: KY-0118

INTERVENTIONS:
Drug: KY-0118 — KY-0118 is to be injected intravenously with a dose of 0.3μg/kg, 1μg/kg, 3μg/kg, 6μg/kg, 12μg/kg, 24μg/kg, 36μg/kg, 48μg/kg or 64μg/kg until disease progresses or unacceptable tolerability occurs;
  Arms: KY-0118
Drug: KY-0118 — KY-0118 is to be injected intravenously with a dose of dose1~dose5 weekly until disease progresses or unacceptable tolerability occurs;
  Arms: Cohort1: KY-0118
Drug: KY-0118 — KY-0118 is to be injected subcutaneously with a dose of dose1~dose5 weekly until disease progresses or unacceptable tolerability occurs;
  Arms: Cohort2: KY-0118

SUMMARY:
This dose escalation and dose expansion study is to evaluate and characterize the tolerability, safety, pharmacokinetics and efficacy profile of single agent KY-0118 in Locally Advanced or Metastatic Solid Tumor Patients.

DETAILED DESCRIPTION:
For Phase Ia It aims to evaluate the safety, tolerability, pharmacokinetic characteristics, pharmacodynamic effect, immunogenicity in subjects with locally advanced or metastatic solid tumor patients , and determine the appropriate dose of KY-0118.

For Phase Ib it aims is to further evaluate the efficacy, safety, tolerability, pharmacokinetic properties, pharmacodynamic effects and immunogenicity of KY-0118 with appropriate dose groups (approximately 3-5 dose groups) in different Administration manner.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old, male or female;
2. Subjects with a documented (histologically- or cytologically-proven) solid tumor malignancy that is locally advanced or metastatic; progression or are intolerant to existing standard therapy or subjects without standard therapy;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；Expected survival time≥ 12 weeks;
4. At least one measurable lesion per RECIST 1.1 (without local treatment or progress after local treatment);
5. Adequate organ function;
6. Toxicity from prior anticancer therapy recovered to ≤ grade 1 prior to the first dose of study drugs;
7. Signed informed consent and willingly adherence to the experimental treatment protocol and visit plan.

Exclusion Criteria:

1. Specific anti-tumor treatment prior to use of study treatment;
2. Immunosuppressants or systemic hormone therapy were being used and were not discontinued within 2 weeks prior to enrollment;
3. IL-2 treatment within 6 months prior to the first dose of study drugs;
4. Any immune related adverse events (irAE) that have occurred during previous immunotherapy medication, with a grade of ≥ 3 or leading to termination of immunotherapy;
5. Primary Central Nervous System (CNS) Malignant Tumors or Active CNS Metastasis with Local Treatment Failure;
6. Any severe and/or uncontrolled diseases, including but not limited to: uncontrolled hypertension or pulmonary hypertension or unstable angina; Chronic heart failure; Valve disease; Severe arrhythmia; Had myocardial infarction or bypass or stent surgery within 6 months before screening;
7. History of arteriovenous thromboembolism within 6 months prior to screening；
8. Moderate or severe respiratory distress at rest due to advanced malignant tumors or their complications or severe primary lung diseases；or a current need for continuous oxygen therapy, or a current history of interstitial lung disease (ILD) or pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc. ;
9. Uncontrolled bleeding or known tendency to bleed; Patients with chronic Crohn's disease and ulcerative colitis;Patients with hereditary nonpolyposis colorectal cancer or familial adenomatous polyposis syndrome;Patients with a history of intestinal perforation and fistula, but not cured after surgical treatment;Esophagogastric varices;
10. Third space effusion that cannot be controlled by puncture and drainage treatment and require repeated drainage or have obvious symptoms;
11. Patients who require extensive fluid replacement assessed by investigators;
12. Active hepatitis B or active hepatitis C;
13. Active infectious process;
14. A history of immunodeficiency;
15. Autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, autoimmune thyroid disease, multiple sclerosis, etc.;
16. Patients with allergic constitution, or known to have a history of allergy to IL-2 or PD-1/PD-L1 drugs or any of their components, or known to have a history of severe allergic reactions to fusion proteins;
17. History of other malignancies within 5 years prior to screening;
18. Surgery (other than diagnostic biopsy) within 4 weeks prior to screening or planned to have surgery during the study period;
19. Had received live vaccine within 4 weeks before the first dose or planned to receive live vaccine during the trial;
20. History of neurological or psychiatric disorders, such as epilepsy, dementia, altered mental status, and poor compliance;
21. History of alcohol or drug abuse within the last 1 year;
22. Women who are pregnant or breastfeeding. Patients unwilling to use a highly effective method of contraception during the study period and for 6 months after receiving the trial drug;
23. Attended other study within 4 weeks prior to screening;
24. Other conditions deemed unsuitable for inclusion by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity (DLT) | 21 days during the first 3-week cycle
Adverse Event | Up to 28 days post last dose
  Incidence of untoward medical occurrences (adverse event = AE) in a participant who received study drug. Adverse events will be evaluated by dosing cohort and recorded according to NCI CTCAE Version 5.0.

SECONDARY OUTCOMES:
Cmax | Up to 7 days post last dose
  Peak expansion
Ctrough | Up to 7 days post last dose
  Trough concentration
Tmax | Up to 7 days post last dose
  time to peak expansion
T1/2 | Up to 7 days post last dose
  Elimination half-life
AUC | Up to 7 days post last dose
  Area under curve
CL | Up to 7 days post last dose
  Clearance rate
Regulatory t cells（Tregs） | Up to 7 days post last dose
  Levels of Tregs in peripheral blood at baseline and during administration;
CD4+ T lymphocyte count | Up to 7 days post last dose
  Levels of CD8+ T lymphocyte count in peripheral blood at baseline and during administration;
CD8+ T lymphocyte count | Up to 7 days post last dose
  Levels of CD8+ T lymphocyte count in peripheral blood at baseline and during administration;
NK cells count | Up to 7 days post last dose
  Levels of NK cells count in peripheral blood at baseline and during administration;
IL-6 | Up to 7 days post last dose
  Levels of IL-6 in peripheral blood at baseline and during administration;
IFN-γ | Up to 7 days post last dose
  Levels of IFN-γ in peripheral blood at baseline and during administration;
TNF-ɑ | Up to 7 days post last dose
  Levels of TNF-ɑ in peripheral blood at baseline and during administration;
Granzyme B | Up to 7 days post last dose
  Levels of Granzyme B in peripheral blood at baseline and during administration;
Perforin | Up to 7 days post last dose
  Levels of perforin in peripheral blood at baseline and during administration;
Objective response rate (ORR) | Up to 28 days post last dose
  To evaluate the preliminary antitumor activity of KY-0118
Progression-free survival (PFS) | Up to 28 days post last dose
  To evaluate the preliminary antitumor activity of KY-0118
Duration of response(DOR) | Up to 28 days post last dose
  To evaluate the preliminary antitumor activity of KY-0118
Disease control rate (DCR) | Up to 28 days post last dose
  To evaluate the preliminary antitumor activity of KY-0118
The incidence of ADA of KY-0118 | Up to 7 days post last dose
  Each subject will be tested for anti-drug (KY-0118) antibody (ADA)
The incidence of NAb of KY-0118 | Up to 7 days post last dose
  Each subject with ADA-positive serum samples will continue to be tested for neutralizing antibodies (NAb)
PD-1 receptor occupancy rate | Up to 7 days post last dose
IL-2 receptor occupancy rate | Up to 7 days post last dose
  IL-2 receptor occupancy of Nk cells, CD8+ T lymphocyte and CD4+T lymphocyte
Ki67 phenotype | Up to 7 days post last dose
  Ki67 phenotype of Nk cells and CD8+T lymphocyte

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - The First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui
  - The Fifth Medical Center of the Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Hubei Province Tumor Hospital, Wuhan, Hubei
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Second People's Hospital of Liaocheng, Liaocheng, Shandong
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Province Tumor Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided